CLINICAL TRIAL: NCT05146011
Title: Clinical Outcomes of Single Stage Versus Two-stage Laparoscopic Roux-en-y Gastric Bypass in the Management of Super Obesity: a Propensity Score Weighted Analysis'
Brief Title: Clinical Outcomes of Single Stage Versus Two-stage Treatment of Severe Obesity
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Principal Investigator, Matyas Fehervari, Honorary Clinical Research Fellow, Imperial College London
Other Study IDs: PCD906
Record Dates: First submitted 2021-11-08; First posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-11

CONDITIONS: Obesity, Morbid
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Single stage pathway
  Interventions: Procedure: Gatsric balloon insertion
- Two stage pathway
  Interventions: Procedure: Gatsric balloon insertion

INTERVENTIONS:
Procedure: Gatsric balloon insertion — Insertion of Gastric balloon prior to laparoscopic gastric bypass surgery

SUMMARY:
Laparoscopic Roux-en-Y gastric bypass (LRYGB) in super obese patients (BMI≥50kg/m2) is a challenging operation. Weight reduction with intragastric balloon (IGB) prior to LRYGB may improve operative outcomes and improves weight loss. We assessed 155 patients, with a BMI≥50 kg/m2 who underwent either intra-gastric balloon (IGB) insertion followed by LRYGB (two-stage group), or LRYGB as the definitive bariatric procedure (single-stage group) in our institution. Two stage procedure was adopted for high-risk individuals.

ELIGIBILITY:
Inclusion Criteria:

* patients, with a BMI≥50 kg/m2, underwent either intra-gastric balloon (IGB) insertion followed by LRYGB (two-stage group), or LRYGB as the definitive bariatric procedure (single-stage group)

Exclusion Criteria:

* NA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients, with a BMI≥50 kg/m2 undergoing Bariatric Surgery in Chelsea and Westminster Hospital
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2000-06 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Percentage of total weight loss measured in kilograms following Bariatric Surgery | 24 months after Bariatric Surgery
  Percentage total weight loss is the proportion of weight lost in kilograms since the intervention of the weight before the intervention. This will be calculated by using the following formula. Initial weight is considered the weight on the day of surgery and Postop weight considered as the weight 24 months following Bariatric Surgery (intervention).
  Percent of total weight loss (%TWL)=((Initial Weight)-(Postop Weight)): Initial Weight x 100
  Weight is expressed in kilograms.
Length of hospital stay in days following Bariatric Surgery | 90 days following gastric bypass surgery
  Hospital stay following laparoscopic gastric bypass surgery measured in days and compared between the groups.

IPD SHARING:
Plan to Share IPD: Undecided